CLINICAL TRIAL: NCT04647877
Title: Enrichment Randomized Double-blind, Placebo-controlled Cross-over Trial With PHEnytoin Cream in Patients With Painful Chronic Idiopathic Axonal polyNEuropathy
Brief Title: Phenytoin Cream for the Treatment of Neuropathic Pain
Acronym: EPHENE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: David J. Kopsky (Other)
Collaborators: Princess Beatrix Muscle Foundation (Other); Dr. C.J. Vaillant Fonds (Unknown)
Responsible Party: Sponsor-Investigator, David J. Kopsky, MD, coordinating researcher, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UMC-NMZ-EPHENE2020
Record Dates: First submitted 2020-11-16; First posted 2020-12-01 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Chronic Idiopathic Axonal Polyneuropathy
Keywords: cryptogenic sensory polyneuropathy; CIAP; neuropathic pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phenytoin 10 percent cream (Experimental): Phenytoin 10 percent cream, 2 to 4 times daily application, 2 weeks long
  Interventions: Drug: phenytoin cream
- Phenytoin 20 percent cream (Experimental): Phenytoin 20 percent cream, 2 to 4 times daily application, 2 weeks long
  Interventions: Drug: phenytoin cream
- Placebo cream (Placebo Comparator): Placebo cream, 2 to 4 times daily application, 2 weeks long
  Interventions: Other: Placebo cream

INTERVENTIONS:
Drug: phenytoin cream — Phenytoin cream to be applied on the neuropathic pain area
  Arms: Phenytoin 10 percent cream; Phenytoin 20 percent cream
Other: Placebo cream — Placebo cream to be applied on the neuropathic pain area
  Arms: Placebo cream

SUMMARY:
Objectives: The main objective is to evaluate the efficacy and safety of phenytoin cream in patients with neuropathic pain due to chronic idiopathic axonal polyneuropathy (CIAP). The second objective is to determine the predictive value of a double-blind placebo-controlled response test (DOBRET) to identify sustained responders.

Study design: This is a 6-week enrichment randomized double-blind, placebo-controlled cross-over trial evaluating phenytoin cream in 84 participants with painful CIAP, whereafter an open label extension phase is offered with phenytoin 20 percent cream for up to one year.

At baseline a DOBRET with phenytoin 10 percent and placebo cream will be performed in each study participant to stratify participants according to their response to the DOBRET before entering the double-blind cross-over phase. DOBRET positive participants are those who experience at least two points pain reduction on the 11-point numerical rating scale (NRS) on the phenytoin 10 percent cream applied area within 30 minutes and at least one-point difference in pain reduction on the NRS between phenytoin 10 percent and placebo cream applied area, in favour of the former.

Participants will receive three treatments in a double blind fashion and in a randomized order: phenytoin 10 percent, phenytoin 20 percent and placebo cream. The duration of each treatment period is two weeks. Participants will cross-over two times to each of the other treatments. The study does not have wash-out periods between treatments, because the mean duration of analgesic effect after an application is expected to be less than nine hours. A blood sample will be collected at the end of the second week of the first treatment period to test for phenytoin plasma levels.

Study population: The investigators aim to include 84 participants, age 40 years or older, who have been diagnoses with painful CIAP at the University Medical Center Utrecht and fulfil the inclusion criteria and have given written informed consent.

Interventions: Phenytoin cream in concentrations of 10 percent and 20 percent cream compared to placebo cream.

Primary endpoint: Change in pain intensity measured on the NRS between baseline and week 2 for phenytoin 20% cream versus placebo cream.

ELIGIBILITY:
Inclusion Criteria:

* Patients have been diagnosed with CIAP defined as: presence of symmetrical distal sensory or sensorimotor symptoms such as numbness, pins and needles, tightness, coldness, unsteadiness, muscle cramps, and weakness with onset in the feet, compatible with polyneuropathy; presence of symmetrical distal sensory or sensorimotor signs with evidence of large nerve fiber involvement such as decreased sense of touch, vibration, and proprioception, usually in the presence of decreased pin prick/temperature sense, decreased/absent tendon reflexes, or slight muscle weakness on neurologic examination, compatible with polyneuropathy; an insidious onset and slow or no progression of the polyneuropathy over the course of at least 6 months; no identifiable cause for the polyneuropathy after thorough history-taking, clinical examination, and extensive laboratory testing; no suggestion of a hereditary polyneuropathy based on detailed kinship history (i.e., one or more affected family member), neurologic examination, or confirmation by genetic analysis; and nerve conduction studies excluding a demyelinating polyneuropathy and confirming large nerve fiber involvement if the findings on neurologic examination are equivocal considering the patient's age.
* Presence of chronic localized neuropathic pain due to CIAP
* Neuropathic pain localized in two anatomically symmetrical areas of feet/lower legs
* Duration of neuropathic pain ≥3 months
* Duration of ≥1 hour neuropathic pain per day
* Neuropathic pain characteristics defined by the Douleur Neuropathique 4 questions (DN4) score ≥4
* Mean pain score during daytime of ≥4 and <10 on the NRS at study entry (baseline)
* Difference of pain intensity between left and right foot and/or lower leg of not more than 1 point on the NRS
* No changes in neuropathic pain medication for at least 1 month
* Absence of any of the exclusion criteria outlined below

Exclusion Criteria:

* Painful (poly)neuropathy other than CIAP
* Presence of neuropathic pain due to any other condition than CIAP
* Neuropathic pain (distribution, duration, characteristics, intensity) not fulfilling the inclusion criteria
* Pregnancy or planned pregnancy in the study period (will only be asked)
* Use of oral phenytoin
* Open wounds in the neuropathic pain area
* Current use of topical analgesics
* Presence of other pain syndromes such as the widespread pain syndrome or pain in joints
* Presence of serious psychological/psychiatric morbidity
* Addiction to intoxicants
* Hypersensitivity to the study medication (active substance and excipients)
* Insufficient mastery of the Dutch language
* Cognitive impairment and insufficiently capable to understand the purpose of the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Change in mean pain intensity measured on the 11-point numerical rating scale (NRS) between baseline and week 2 for phenytoin 20% cream versus placebo cream. | Mean baseline vs. mean of second week of each intervention
  0 = no pain, 10 = worst imaginable pain. The bigger the mean change, the better the outcome

SECONDARY OUTCOMES:
Change in mean pain intensity from baseline 11-point numerical rating scale (NRS) to the mean NRS in the second week in double-blind response test in positive and negative participants and all participants combined | Mean baseline vs. mean of second week of each intervention
  0 = no pain, 10 = worst imaginable pain. The bigger the mean change, the better the outcome
Change of EuroQol (EQ5-5D-5L) from baseline to the end of the second week of each treatment period | Baseline vs. end of second week of each intervention
  EQ5-5D-5L consists of 5 quality of life questions assessed on a 5 point scale: the lower the score, the better quality of life. Furthermore, a visual analogue scale from 0 to 100 is included. The higher the score, the better quality of life.
Change of Neuropathic Pain Symptom Inventory (NPSI) from baseline to the end of the second week of each treatment period | Baseline vs. end of second week of each intervention
  The NPSI consists of 10 neuropathic pain descriptors on the NRS, and 2 items assessing the duration of spontaneous ongoing and paroxysmal pain. The lower the score, the less pain.
Change of subscales of the Brief Pain Inventory (sBPI) from baseline to the end of the second week of each treatment period | Baseline vs. end of second week of each intervention
  The sBPI consists of 7 quality of life questions, assessed on the NRS. The lower the score, the better quality of life.
Change of the 3 worst pain characteristics from baseline to the end of the second week of each treatment period | Baseline vs. end of second week of each intervention
  The 3 worst pain characteristics are scored on the NRS. The lower the score, the less pain.
Change of Patient Global Impression of Change Scale (PGIC) from baseline to the end of the second week of each treatment period | Baseline vs. end of second week of each intervention
  The PGIC is a 7-point satisfaction scale. The lower the score, the better.
30 percent and 50 percent improvement or more on the NRS compared to placebo within one patient | Baseline vs. end of second week of each intervention
Time of carry-over effects after a treatment period | First week of each intervention
Onset of analgesic effect after application | At the end of second week of each intervention
  The onset of analgesic effect will be noted in minutes.
Duration of analgesic effect | At the end of second week of each intervention
  The duration of analgesic effect will be noted in hours.
Daily number of cream applications | At the end of second week of each intervention
Percentage of analgesic effect as rated by the participant | At the end of second week of each intervention.
  The participant will be asked about the percentage of pain reduction at the end of the second week of each intervention. The higher, the better.
Local and/or systemic side effects | During the 6 weeks of double-blind phase and 1 year open phase
  At each visit and telephone call participants will be asked about possibly occurring side effects.
Detection of phenytoin in plasma | At the end of second week of first treatment period
  Two hours after last application phenytoin plasma level will be evaluated
Predictive value of DOBRET | Baseline vs. mean of second week of each intervention
  Correlation with DOBRET response and mean pain reduction while using phenytoin 10 percent or 20 percent cream. The stronger the correlation, the more predictive the DOBRET is.
Use of escape pain medication | During the 6 weeks of double-blind phase and 1 year open phase
  The daily amount of acetaminophen and/or non-steroid anti-inflammatory drugs

CONTACTS AND LOCATIONS:
Overall Officials: Alexander FJE Vrancken, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kopsky DJ, Vrancken AFJE, Keppel Hesselink JM, van Eijk RPA, Notermans NC. Usefulness of a Double-Blind Placebo-Controlled Response Test to Demonstrate Rapid Onset Analgesia with Phenytoin 10% Cream in Polyneuropathy. J Pain Res. 2020 May 1;13:877-882. doi: 10.2147/JPR.S243434. eCollection 2020. PMID 32431536
- [Background] Kopsky DJ, Keppel Hesselink JM. Single-Blind Placebo-Controlled Response Test with Phenytoin 10% Cream in Neuropathic Pain Patients. Pharmaceuticals (Basel). 2018 Nov 12;11(4):122. doi: 10.3390/ph11040122. PMID 30424471
- [Background] Kopsky DJ, Keppel Hesselink JM. Phenytoin Cream for the Treatment for Neuropathic Pain: Case Series. Pharmaceuticals (Basel). 2018 May 28;11(2):53. doi: 10.3390/ph11020053. PMID 29843362
- [Background] Kopsky DJ, Keppel Hesselink JM, Russell AL, Vrancken AFJE. No Detectable Phenytoin Plasma Levels After Topical Phenytoin Cream Application in Chronic Pain: Inferences for Mechanisms of Action. J Pain Res. 2022 Feb 9;15:377-383. doi: 10.2147/JPR.S345347. eCollection 2022. PMID 35173477
- [Derived] Kopsky DJ, van Eijk RPA, Warendorf JK, Keppel Hesselink JM, Notermans NC, Vrancken AFJE. Enriched enrollment randomized double-blind placebo-controlled cross-over trial with phenytoin cream in painful chronic idiopathic axonal polyneuropathy (EPHENE): a study protocol. Trials. 2022 Oct 22;23(1):888. doi: 10.1186/s13063-022-06806-8. PMID 36273216
- See also: Related Info — http://www.topicalinnovations.com